CLINICAL TRIAL: NCT00706290
Title: Brief CBT for Anxiety and Advanced Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joseph A. Greer, Ph.D., Clinical Assistant in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CDR0000597438; 1R03CA128478-01 (NIH); 2007P000368 (Other: Partners Human Research Committee Protocol Number)
Record Dates: First submitted 2008-06-26; First posted 2008-06-27 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety; Depression; Unspecified Adult Solid Tumor, Protocol Specific; Cancer; Cognitive Behavioral Therapy
Keywords: anxiety; depression; quality of life; psychosocial effects of cancer and its treatment; advanced cancer; metastatic cancer; stage IV cancer; cognitive behavioral therapy
MeSH Terms: conditions — Anxiety Disorders; Depression; Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention - CBT (Experimental): Participants randomized to the intervention group received cognitive behavioral therapy (CBT) for anxiety after completing a baseline assessment consisting of clinician administered psychiatric evaluations and a psychosocial self-report battery. After completing the CBT intervention, consisting of 6-7 sessions over the course of 2-3 months, participants completed a post-intervention assessment identical to the baseline.
  Interventions: Behavioral: Brief Cognitive Behavioral Therapy
- Routine Care Control (No Intervention): Participants randomized to the control condition completed a baseline assessment consisting of clinician administered psychiatric evaluations and a psychosocial self-report battery. They then received routine medical care. After 2 months and after completing the post clinical assessment identical to the baseline, they were offered the opportunity to receive the CBT intervention for free. This ensured that all participants ultimately received cognitive-behavioral therapy if desired, while permitting an examination of the effect size for the intervention compared to routine care.

INTERVENTIONS:
Behavioral: Brief Cognitive Behavioral Therapy — The cognitive-behavioral intervention consists of 6-7 sessions lasting 60-90 minutes each focused on psycho-education; relaxation training; cognitive-restructuring and coping with cancer fears; and activity planning and pacing. Sessions are delivered by a licensed clinical psychologist or trained psychology fellow or graduate student.
  Other Names: Brief CBT; CBT
  Arms: Intervention - CBT

SUMMARY:
RATIONALE: Providing cognitive-behavioral therapy (CBT) may reduce anxiety and improve quality of life of patients with advanced cancer.

PURPOSE: To examine the development and pilot testing of a brief cognitive-behavioral therapy intervention to treat anxiety and improve quality of life in patients with advanced cancer.

Hypothesis: Patients with anxiety associated with advanced cancer who receive CBT will report significantly fewer anxiety symptoms compared to those in the comparison condition.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop and examine the feasibility and patient acceptability of administering a manualized cognitive-behavioral intervention that improves quality of life by treating anxiety in patients with advanced cancer.
* To estimate the effect size of a manualized cognitive-behavioral intervention to reduce anxiety in patients with advanced cancer.
* To estimate the effect size for the secondary outcomes (i.e., depression and quality of life) and to examine the extent to which specific variables (i.e., sex, age, chemotherapy side effects, pain levels) are consistent with the conceptual model as potential moderators of treatment effect.

OUTLINE: This is a pilot study followed by a randomized study. Patients are stratified according to type of cancer.

* Pilot study: Patients complete qualitative interviews to explore ways that anxiety impacts patients, to identify components of a cognitive-behavioral therapy intervention that are most useful, and to determine the optimal method of delivery for the intervention (e.g., number and timing of interventions, administration during chemotherapy infusions when feasible). Based upon these results a full treatment manual is written for use in the randomized study.

Patients are then randomized to 1 of 2 treatment arms.

* Arm I (cognitive-behavioral therapy): Patients undergo six-seven 90-minute treatment sessions (over 2 months) based on the results of the pilot study. Modules include psychoeducation and goal setting; relaxation training; cognitive restructuring; coping with cancer fears; activity planning and pacing; and review, termination, and plan for continued use of skills.
* Arm II (routine care): Patients receive routine medical care.

At the completion of treatment, all participants meet with a blinded independent assessor to assess outcomes. Patients undergo psychiatric evaluation, including the Hamilton Anxiety Rating Scale (HAM-A), the Montgomery Asberg Depression Rating Scale (MADRS), the Mini International Neuropsychiatric Interview (MINI), and a psychosocial self-reported battery at baseline and after 2-3 months.

After completing treatment, patients who underwent routine care (arm II) may undergo cognitive-behavioral therapy as in arm I, if desired.

ELIGIBILITY:
INCLUSION CRITERIA:

* Diagnosis of incurable solid tumor cancers
* At least four weeks post-diagnosis
* Current symptoms of anxiety and anxiety as principal psychiatric problem

  * Patients with co-morbid depression are eligible as long as anxiety symptoms are primary
  * Concurrent pharmacotherapy for anxiety allowed

EXCLUSION CRITERIA:

* Delirium or dementia
* Active and untreated major psychiatric condition such as schizophrenia or bipolar disorder, other psychotic disorders, or substance dependence
* Other inability to complete informed consent process or study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-04; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms as measured by the Hamilton Anxiety Rating Scale | 1) At enrollment pre-intervention. 2) Post intervention (2-3 months after enrollment)
  The Hamilton Anxiety Ratings Scale (HAM-A) consists of 14 items that provide an overall measure of global anxiety.

SECONDARY OUTCOMES:
Depression as measured by the Montgomery Asberg Depression Rating Scale | 1) At enrollment pre-intervention. 2) Post intervention (2-3 months after enrollment)
  The Montgomery Asberg Depression Rating Scale (MADRS) is an empirically derived 10-item interview that measures depression symptoms.
Quality of life as measured by the Functional Assessment of Scale Cancer Therapy (FACT-G) | 1) At enrollment pre-intervention. 2) Post intervention (2-3 months after enrollment)
  Consisting of 28 items, the FACT-G has four subscales assessing physical, functional, emotional, and social well-being during the past 7 days. Higher scores on the total score and each subscale indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Greer, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Greer JA, Traeger L, Bemis H, Solis J, Hendriksen ES, Park ER, Pirl WF, Temel JS, Prigerson HG, Safren SA. A pilot randomized controlled trial of brief cognitive-behavioral therapy for anxiety in patients with terminal cancer. Oncologist. 2012;17(10):1337-45. doi: 10.1634/theoncologist.2012-0041. Epub 2012 Jun 11. PMID 22688670
- [Result] Greer JA, Park ER, Prigerson HG, Safren SA. Tailoring Cognitive-Behavioral Therapy to Treat Anxiety Comorbid with Advanced Cancer. J Cogn Psychother. 2010 Jan 1;24(4):294-313. doi: 10.1891/0889-8391.24.4.294. PMID 21234281